CLINICAL TRIAL: NCT02356003
Title: TICS: Transcranial Magnetic Stimulation for Children With Tourette's Syndrome
Brief Title: Transcranial Magnetic Stimulation for Children With Tourette's Syndrome
Acronym: TICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Frank MacMaster, PhD, Assistant Professor, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB14-1839
Record Dates: First submitted 2015-01-31; First posted 2015-02-04 (Estimated); Results first posted 2020-04-13 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Tourette Syndrome
Keywords: Tourette Syndrome; Children; Tics
MeSH Terms: conditions — Tourette Syndrome; Tics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low frequency rTMS (Experimental): Eleven children (7-12 years of age) with Tourette syndrome will be undergo low frequency repetitive transcranial magnetic stimulation (5 times a week for three weeks).
  Interventions: Device: Low frequency repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Low frequency repetitive transcranial magnetic stimulation — Baseline high-resolution anatomical magnetic resonance images will allow individualized neuronavigation (Brainsight 2, Rogue Research, Montreal QC) to co-register the transcranial magnetic stimulation Airfilm coil (Magistim, UK) precisely to the supplementary motor area as defined by functional magnetic resonance imaging. Interventional low frequency repetitive transcranial magnetic stimulation parameters will be: intensity 100% resting motor threshold, frequency 1 Hz, duration = 20 minutes (1200 stimulations). Treatments will occur on each weekday at the same time of day for three weeks (15 total). These are standard parameters for low frequency repetitive transcranial magnetic stimulation and are well tolerated in children.

SUMMARY:
Tics are the core symptom of Tourette syndrome. These are repetitive, sudden, semi-voluntary movements or sounds. In some children, these tics can be especially bad and require treatment, however, options are limited. It is only with time and practice that youth with Tourette syndrome are better able to suppress their tics. For these reasons, new interventions are needed. The investigators will target a brain region involved in tics called the supplementary motor area. Using low frequency repetitive transcranial magnetic stimulation, the investigators will inhibit the activity, in a similar way to the tic suppression that develops with age. The investigators propose the following objectives: (Aim 1) The investigators hypothesize that Tourette syndrome symptom severity (as measured by the Yale Global Tic severity Scale) will decrease with low frequency repetitive transcranial magnetic stimulation targeting the supplementary motor area. (Aim 2) The investigators further hypothesize that improvement in Tourette syndrome symptoms will be moderated by low frequency repetitive transcranial magnetic stimulation induced changes in GABA and glutamate in the supplementary motor area, and changes in the functional connectivity between the supplementary motor area and primary motor cortex. Eleven children (7-12 years of age) with Tourette syndrome will be undergo low frequency repetitive transcranial magnetic stimulation (five times a week for three weeks). After the three weeks, they will look for changes in tic severity and brain chemistry and function. By developing a novel avenue for treating Tourette syndrome, they can directly impact the care of children by reducing the severity of tics and improving quality of life.

DETAILED DESCRIPTION:
Background Tourette syndrome is very common. It affects over 80,000 Canadian youth. Tics are the core symptom of Tourette syndrome. These are repetitive, sudden, semi-voluntary movements or sounds. In some children, these tics can be especially bad and require treatment, however, options are limited. Medications for Tourette syndrome carry significant risk of side effects. Behavioral treatments, like habit reversal therapy, show promise and are safe, but are difficult to apply to younger children. It is only with time and practice that youth with Tourette syndrome are better able to suppress their tics. Finally, neither medication nor behavior therapies directly target the root cause of the tics. For these reasons, new interventions are needed.

Specific Objectives The investigators will target a key brain region involved in tics. It is called the supplementary motor area. Using low frequency repetitive transcranial magnetic stimulation, they will inhibit the activity of that brain region, in a similar way to the tic suppression that develops with age.

The investigators propose the following specific objectives:

(Aim 1) The investigators will characterize the effect of low frequency repetitive transcranial magnetic stimulation of the supplementary motor area on Tourette syndrome symptoms. They hypothesize that Tourette syndrome symptom severity (as measured by the Yale Global Tic severity Scale) will decrease with low frequency repetitive transcranial magnetic stimulation targeting the supplementary motor area.

(Aim 2) The investigators will identify the changes in brain metabolites (glutamate and GABA) and functional connectivity caused by low frequency repetitive transcranial magnetic stimulation that normalize brain activity. They hypothesize that improvement in Tourette syndrome symptoms will be moderated by low frequency repetitive transcranial magnetic stimulation induced changes in GABA and glutamate in the supplementary motor area. This will be assessed with proton magnetic resonance spectroscopy, potentiation of GABAergic neurotransmission assessed with short-interval cortical inhibition, and changes in the functional connectivity between the supplementary motor area and primary motor cortex.

Methods Eleven children (7-12 years of age) with Tourette syndrome will be undergo low frequency repetitive transcranial magnetic stimulation (5 times a week for three weeks). The investigators will assess the key variables with interviews and brain imaging of the children before and after the three-week intervention. After the three weeks, they will look for changes in tic severity and brain chemistry and function.

Expected Results The investigators have pioneered transcranial magnetic stimulation applications in child and adolescent populations. By developing a novel avenue for treating Tourette syndrome, they can directly impact the care of children by reducing the severity of tics and improving quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Right-handed

Exclusion Criteria:

* Female
* Left-handed
* Comorbid Attention Deficit Hyperactivity Disorder

Ages: 7 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank p MacMaster, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Frequency rTMS: Ten children (7-12 years of age) with Tourette syndrome will be undergo low frequency repetitive transcranial magnetic stimulation (5 times a week for three weeks).
  Low frequency repetitive transcranial magnetic stimulation: Baseline high-resolution anatomical magnetic resonance images will allow individualized neuronavigation (Brainsight 2, Rogue Research, Montreal QC) to co-register the transcranial magnetic stimulation Airfilm coil (Magistim, UK) precisely to the supplementary motor area as defined by functional magnetic resonance imaging. Interventional low frequency repetitive transcranial magnetic stimulation parameters will be: intensity 100% resting motor threshold, frequency 1 Hz, duration = 20 minutes (1200 stimulations). Treatments will occur on each weekday at the same time of day for three weeks (15 total). These are standard parameters for low frequency repetitive transcranial magnetic stimulation and are well tolerated in children.
Period: Overall Study
Arm/Group | Low Frequency rTMS
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Low Frequency rTMS
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.524 (1.995)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 10
Yale Global Tic Severity Scale (YGTSS) [Mean (Standard Deviation); unit: units on a scale] — The Yale Global Tic Severity Scale (YGTSS) quantifies the severity of tic symptoms in individuals aged 6-17 years. The YGTSS is a semi-structured interview where individuals are asked to rate the severity of their tic symptoms (motor and vocal; number, frequency, intensity, complexity, and interference). There is also an impairment scale, where the participant rates how tics impact their daily life. The Total Tic Severity Score has a range of 0-50, and the Global Severity Score has a range of 0- 100. A higher score on all scales suggests greater tic severity.
  units on a scale | 64.40 (19.83)

OUTCOME MEASURES:

1. Primary Outcome: Yale Global Tic Severity Scale
Description: Measure of tic severity using the Yale Global Tic Severity Scale (YGTSS). This is the standard measure for studies of Tourette's syndrome. The Global Severity Score has a range of 0- 100. A higher score on all scales suggests greater severity of tics.
Time Frame: Four weeks
Population: We stopped recruitment at 10 as the study ran out of money.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Frequency rTMS
Number analyzed (Participants) | 10
units on a scale
  Baseline | 64.40 (19.83)
  Post-rTMS | 26.40 (14.86)

2. Secondary Outcome: Glutamate Concentration
Description: Glutamate concentration in the supplementary motor area
Time Frame: Four weeks
Population: We stopped recruitment at 10 as the study ran out of money.
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | Low Frequency rTMS
Number analyzed (Participants) | 10
mM
  Baseline | 14.2 (1.73)
  Post-rTMS | 13.4 (1.38)

3. Secondary Outcome: Functional Connectivity
Description: Functional connectivity between the supplementary motor area and primary motor cortex as measured with resting state functional magnetic resonance imaging (rs-fMRI). T-value is the fMRI statistic that shows the level of connectivity. The higher the T-value, the greater the level of connectivity.
Time Frame: Four weeks
Measure: Number; unit: T-value
Arm/Group | Low Frequency rTMS
Number analyzed (Participants) | 10
T-value | 1.89

ADVERSE EVENTS:
Time Frame: The three weeks of the intervention and the week following.
Description: We have a scale for tolerability and adverse events that we use for all TMS studies.
Arm/Group | Low Frequency rTMS
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
This was a pilot open label trial of rTMS and as such subject to the standard limitations of all pilot intervention studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT02356003/Prot_SAP_000.pdf